CLINICAL TRIAL: NCT04094844
Title: A Randomized Trial of Roadmap 2.0
Brief Title: Health Information Technology System ("Roadmap 2.0") in the Context of Hematopoietic Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2019.106; HUM00165192 (Other: University of Michigan); HUM00186436 (Other: University of Michigan); R01HL146354 (NIH)
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Hematologic Diseases
Keywords: Hematopoietic Cell Transplantation; Mobile Health Technology
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Intervention Model Description: * Active comparator arm: Adult caregivers (n=166) with adult patients >/= 18 years of age (n=83) and pediatric patient <18 years of age (n=83)
  * Experimental arm: Adult caregivers (n=166) with adult patients >/= 18 years of age (n=83) and pediatric patient <18 years of age (n=83)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roadmap 2.0 (Active Comparator): Roadmap 2.0 mobile app + wearable sensor to track activity and sleep + usual care (informational or educational resources provided through verbal communication or written hand-out materials).
  Includes caregivers of adult patients and caregivers of pediatric patients
  Interventions: Other: Wearable activity sensor; Behavioral: Roadmap 2.0 information system; Other: Survey administration
- Roadmap 2.0 with Positive Activities (Experimental): Roadmap 2.0 mobile app (patients), Roadmap 2.0 with mobile Positive Activities app (caregivers) + wearable sensor to track activity and sleep + usual care (informational or educational resources provided through verbal communication or written hand-out materials).
  Includes caregivers of adult patients and caregivers of pediatric patients
  Interventions: Other: Wearable activity sensor; Other: Survey administration; Behavioral: Roadmap 2.0 information system with Positive Activities

INTERVENTIONS:
Other: Wearable activity sensor — Caregivers and patients in both arms of the study will have a Fitbit wearable activity sensor to track activity and sleep.
  Other Names: Fitbit Charge 3
Behavioral: Roadmap 2.0 information system — Caregivers and patients download the Roadmap 2.0 app on their mobile phones or tablets
  Arms: Roadmap 2.0
Other: Survey administration — Caregivers and patients will be asked to respond to survey questions at 3 timepoints.
  Other Names: PROMIS®
Behavioral: Roadmap 2.0 information system with Positive Activities — Caregivers and patients download the Roadmap 2.0 app on their mobile phones. Caregivers and patients will be instructed on how to operate Roadmap 1.0 on an iPad (inpatient only) and Roadmap 2.0 on a mobile phone (inpatient and outpatient). Caregivers download the Positive Activities app onto their mobile phone to use freely throughout inpatient and outpatient (through day 120 post-transplant). Caregiver may also use an electronic tablet provided by the study team during the patient's hospital stay.
  Arms: Roadmap 2.0 with Positive Activities

SUMMARY:
The purpose of this research study is to measure the effects of using a mobile phone app (Roadmap 2.0) on the health-related quality of life of caregivers and patients undergoing allogeneic/autologous hematopoietic cell transplantation (HCT).

DETAILED DESCRIPTION:
Health information technology tools may enable caregivers and patients to become more active participants in their healthcare.This study is not to provide any treatment, but rather to investigate the use of this mobile health technology-mediated intervention (Roadmap 2.0). Roadmap 2.0 is a web-based application that integrates patient-specific information and includes several domains: laboratory results, medications, clinical trial details, photos of the healthcare team, trajectory of transplant process, and discharge checklist.

This trial is anticipated to enroll 664 participants, but only caregivers (332 total) will be evaluated for the primary and secondary outcome measures. Thus, the sample size is 332. The total enrollment includes 166 caregiver-patient dyads of adult patients (age >/=18 years) undergoing HCT ("adult dyads" = 332 total) and 166 caregiver-patient dyads of pediatric patients (age 5-17 years) undergoing HCT ("pediatric dyads" = 332 total).

ELIGIBILITY:
Inclusion Criteria

* The caregiver must have an eligible patient (see below)
* The caregiver must be of age ≥18 years.
* The caregiver should be comfortable in reading and speaking English and signing informed consents.
* The caregiver should provide at least 50% of care needs.
* An eligible patient is one who identifies the eligible caregiver as their primary caregiver (i.e., provides at least 50% of care needs).
* An eligible patient is age ≥5 years.
* An eligible patient is scheduled to undergo HCT.
* An eligible patient is able to sign informed consent/assent forms.
* Patients and caregivers agree to provide informed consent that is in regulatory compliance and IRBMED-approved and also in accordance to institutional guidelines. A patient is able to undergo HCT at the U-M only if a designated family caregiver (e.g., parents, adult children, spouses, family members, neighbors, friends) accepts the roles, in accordance to the Clinical Practice Guidelines of the U-M BMT Program.
* The caregiver and patient must have his/her own smartphone to participate.

Exclusion Criteria

- Patient does not meet eligibility criteria to undergo HCT at the U-M BMT Program or Oregon Health & Sciences University.

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2024-08-11 (Actual); Study Completion 2024-08-11 (Actual)

PRIMARY OUTCOMES:
Caregiver health-related quality of life (HRQOL) assessed by the PROMIS Global Health scale. | At day 120 post-transplant
  Mean Global Health scores for each arm at day 120. PROMIS® instruments are scored using item-level calibrations. This method of scoring uses "response pattern scoring," which uses responses to each item for each participant.

OTHER OUTCOMES:
Caregiver health-related quality of life (HRQOL) assessed by PROMIS Profile 29+2 (exploratory) | At day 120 post-transplant
  Mean Profile 29+2 scores for each arm at day 120. PROMIS® instruments are scored using item-level calibrations. This method of scoring uses "response pattern scoring," which uses responses to each item for each participant. This is an exploratory measure.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Won Choi, MD, MS, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cao X, Rozwadowski M, Braun TM, Carlozzi NE, Hassett AL, Johnson AK, Shereck E, Hanauer DA, Choi SW. A Mobile Health Intervention in Caregivers of Patients Undergoing Hematopoietic Cell Transplantation: A Randomized Controlled Trial to Examine Health-Related Quality of Life. BMC Digit Health. 2025;3(1):22. doi: 10.1186/s44247-025-00165-5. Epub 2025 Jul 15. PMID 40822733
- [Derived] Caparso C, Ozkan G, Kluge M, Salim H, Khaghany A, Blok A, Choi SW. Mobile Technology to Monitor and Support Health and Well-Being: Qualitative Study of Perspectives and Design Suggestions From Patients Undergoing Hematopoietic Cell Transplantation. JMIR Form Res. 2023 Aug 31;7:e49806. doi: 10.2196/49806. PMID 37651172
- [Derived] Rozwadowski M, Dittakavi M, Mazzoli A, Hassett AL, Braun T, Barton DL, Carlozzi N, Sen S, Tewari M, Hanauer DA, Choi SW. Promoting Health and Well-Being Through Mobile Health Technology (Roadmap 2.0) in Family Caregivers and Patients Undergoing Hematopoietic Stem Cell Transplantation: Protocol for the Development of a Mobile Randomized Controlled Trial. JMIR Res Protoc. 2020 Sep 18;9(9):e19288. doi: 10.2196/19288. PMID 32945777